CLINICAL TRIAL: NCT03457116
Title: Narcotics vs Non-steroidal Ant Inflammatory Drugs Post-operative Analgesia in Outpatient Rhinoplasty
Brief Title: Narcotics vs NSAIDs for Post-operative Analgesia in Outpatient Rhinoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01839
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Rhinoplasty; Non-steroidal Ant Inflammatory Drugs; Opioid Use
MeSH Terms: interventions — oxycodone-acetaminophen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSAIDS (Active Comparator): 400mg of Ibuprofen
  Interventions: Drug: NSAID
- Opiates (Active Comparator): Norco (hydrocodone 5mg- acetaminophen 325mg)
  Interventions: Drug: Norco

INTERVENTIONS:
Drug: Norco — 20 tablets of Hydrocodone 5mg-Acetaminophen 325mg (Norco)
  Arms: Opiates
Drug: NSAID — Ibuprofen 400mg for post-operative pain
  Arms: NSAIDS

SUMMARY:
The purpose of this study is to compare the efficacy and safety of oral opiate pain medication vs non-steroidal ant inflammatory drugs (NSAIDs) in the treatment of postoperative rhinoplasty pain. This study will also evaluate potential contributing factors affecting the efficacy of these pain control methods. Patients will be randomized to receive either NSAIDs in the form of 400mg of Ibuprofen or Norco (hydrocodone 5mg- acetaminophen 325mg) to be used for post-operative pain. The study will then compare which is more effective in controlling post operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years old undergoing septorhinoplasty or rhinoplasty for either obstructive or aesthetic reasons. All approaches to rhinoplasty and surgical techniques utilized will be included. This will include patients that undergo additional procedures during the rhinoplasty including osteotomies, turbinate reduction, septoplasty, nasal valve repair and ear cartilage graft.

Exclusion Criteria:

* Patients who undergo a rhinoplasty requiring a rib cartilage graft for the procedure as this is known to cause significant pleuritic chest pain.
* Patients receiving functional endoscopic sinus surgery concurrently with the rhinoplasty will be excluded.
* Patients with known history of gastrointestinal bleeds, peptic ulcer disease or who have other comorbidities that prevent them from taking NSAIDs.
* Patients with a history of radiation, active head and neck malignancy or other pain disorders such as various rheumatologic diseases will be excluded to decrease confounding factors in the control of pain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Lee, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Data are available indefinitely at (Link to be included).
Access Criteria: Anyone who wishes to access the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NSAIDS | Opiates
Started | 41 | 29
Completed | 41 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NSAIDS | Opiates | Total
Number analyzed (Participants) | 41 | 29 | 70
Age, Continuous [Mean (Full Range); unit: years] | 32 [19 to 70] | 32 [21 to 64] | 32 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 22 | 17 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 41 | 29 | 70

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Score
Description: Pain scores are reported via Post-Operative Pain Management Survey. On a scale of 1-10, participants indicate how much pain they were in on their pain regiment. The higher the score, the worse the pain (1 = no pain, 10 = worst pain possible)
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NSAIDS | Opiates
Number analyzed (Participants) | 41 | 29
score on a scale | 2.54 (1.57) | 3.14 (1.75)

2. Primary Outcome: Average Pain Score
Description: as for outcome 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NSAIDS | Opiates
Number analyzed (Participants) | 41 | 29
score on a scale | 1.84 (1.29) | 2.46 (1.90)

3. Primary Outcome: Average Pain Score
Description: as for outcome 1
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NSAIDS | Opiates
Number analyzed (Participants) | 41 | 29
score on a scale | 3.29 (2.14) | 3.14 (2.12)

4. Primary Outcome: Average Post-Operative Day (POD) of Medication Cessation
Description: Self-reported via Post-Operative Pain Management Survey
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NSAIDS | Opiates
Number analyzed (Participants) | 41 | 29
days | 4.73 (1.57) | 4.28 (2.23)

5. Secondary Outcome: Number of Participants in NSAIDs Group Who Were Upgraded to Opiates Due to High Levels of Pain
Time Frame: Day 7
Population: This outcome measure is only applicable to NSAIDS
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDS
Number analyzed (Participants) | 41
Participants | 5

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | NSAIDS | Opiates
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/29
Other Adverse Events (participants affected / at risk) | 0/41 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03457116/Prot_SAP_000.pdf